CLINICAL TRIAL: NCT05781802
Title: Assessment of V/Q Matching During Pressure Support Ventilation With Electrical Impedance Tomography
Brief Title: V/Q Matching in Pressure Support Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Andrea Cortegiani, MD, Clinical Professor, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Other Study IDs: EIT01
Record Dates: First submitted 2023-02-27; First posted 2023-03-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Failure; ARDS; Electrical Impedance Tomography
Keywords: Electrical impedance tomography; ARDS; V/Q matching

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult mechanically ventilated patients with ARDS: Adult mechanically ventilated patients with ARDS (see inclusion/exclusion criteria)
  Interventions: Other: Level of pressure support

INTERVENTIONS:
Other: Level of pressure support — Patients will be evaluated in two different conditions sequentially. The first condition will be at a clinically selected level of pressure support under stable clinical conditions.
  This condition will be labeled according to P0.1:
  * In case of P0.1<2, the clinically selected level of pressure support will be considered "High Pressure support".
  * In case of P0.1>2, the clinically selected level of pressure support will be considered "Low Pressure support".
  After data collection at clinically selected level of pressure support, pressure support level will be transiently increased or decreased (i.e. from high to low/ from low to high) to the lowest/highest clinically tolerated level, aiming at the predefined P01 thresholds, and then kept for 20 minutes under stable clinical conditions. Data collection will be repeated and then the clinically selected level of pressure support restored.

SUMMARY:
The aim of this study is to describe the effects of different levels of pressure support on ventilation-perfusion matching in patients recovering from ARDS, using electrical impedance tomography.

DETAILED DESCRIPTION:
Spontaneous breathing during mechanical ventilation has been attributed to both protective and negative effects on patient outcomes, largely varying based on the severity of lung injury. Indeed, in severe ARDS the avoidance of spontaneous efforts has an established protective role. However, spontaneous breathing promotes the distribution of tidal volume towards the dependent lung, and low levels of support pressure determine more homogeneous ventilation in patients recovering from ARDS, compared to higher support levels. Physiology supports the potential of spontaneous breathing to increase lung perfusion, through the decrease of intra-thoracic pressure leading to an increased venous return. This mechanism, in absence of right ventricular dysfunction, may lead to increased global lung perfusion. Furthermore, gas exchange improvements in experimental lung injury models during pressure support vs. controlled ventilation have been explained with redistribution of lung perfusion to nondependent lung areas and improvement of V/Q matching even in absence of significant lung recruitment.

Electrical impedance tomography has been clinically used as a non-invasive tool to assess V/Q matching in patients with ARDS and to compare V/Q matching prior to and after a cycle of prone position in spontaneously breathing patients with COVID-19.

The aim of this study is to describe the effects of different levels of pressure support on ventilation-perfusion matching in patients recovering from ARDS, using electrical impedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Need for invasive mechanical ventilation and ICU admission
* Diagnosis of ARDS at ICU admission or during ICU stay
* Informed consent
* Presence of central line in the internal jugular vein

Exclusion Criteria:

* Any contraindication to Electrical impedance tomography monitoring (e. g. severe chest trauma or wounds)
* Cardiogenic pulmonary edema
* Pulmonary embolism
* Chronic obstructive pulmonary disease
* Pulmonary fibrosis
* Asthma exacerbation
* Pneumothorax and/or chest drainages
* Pre-existing diaphragmatic function impairment
* Neuro-muscular disease or impairment
* Moribund patients with limitation of care or expected survival <48h according to the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were admitted to ICU with acute respiratory distress syndrome (ARDS) or developing it during ICU stay.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in ventilation-perfusion matching | Measured after at least 20 minutes from the application of each of the levels of pressure support and at clinical stability
  Changes in ventilation-perfusion matching between the two different levels of pressure support ("high" level of pressure support and "low" level of pressure support)

SECONDARY OUTCOMES:
Changes in gas exchange | Measured after at least 20 minutes from the application of each of the levels of pressure support and at clinical stability
  Changes in gas exchange measured by blood gas analysis between the two different levels of pressure support ("high" level of pressure support and "low" level of pressure support)
Changes in regional ventilation distribution | Measured after at least 20 minutes from the application of each of the levels of pressure support and at clinical stability
  Changes in regional ventilation distribution between the two different levels of pressure support ("high" level of pressure support and "low" level of pressure support)
Changes in regional perfusion distribution | Measured after at least 20 minutes from the application of each of the levels of pressure support and at clinical stability
  Changes in regional perfusion distribution between the two different levels of pressure support ("high" level of pressure support and "low" level of pressure support)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone. Università degli Studi di Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] Wrigge H, Zinserling J, Neumann P, Defosse J, Magnusson A, Putensen C, Hedenstierna G. Spontaneous breathing improves lung aeration in oleic acid-induced lung injury. Anesthesiology. 2003 Aug;99(2):376-84. doi: 10.1097/00000542-200308000-00019. PMID 12883410
- [Background] Mauri T, Bellani G, Confalonieri A, Tagliabue P, Turella M, Coppadoro A, Citerio G, Patroniti N, Pesenti A. Topographic distribution of tidal ventilation in acute respiratory distress syndrome: effects of positive end-expiratory pressure and pressure support. Crit Care Med. 2013 Jul;41(7):1664-73. doi: 10.1097/CCM.0b013e318287f6e7. PMID 23507723
- [Background] Carvalho AR, Spieth PM, Guldner A, Cuevas M, Carvalho NC, Beda A, Spieth S, Stroczynski C, Wiedemann B, Koch T, Pelosi P, de Abreu MG. Distribution of regional lung aeration and perfusion during conventional and noisy pressure support ventilation in experimental lung injury. J Appl Physiol (1985). 2011 Apr;110(4):1083-92. doi: 10.1152/japplphysiol.00804.2010. Epub 2011 Jan 26. PMID 21270348
- [Background] Carvalho AR, Spieth PM, Pelosi P, Beda A, Lopes AJ, Neykova B, Heller AR, Koch T, Gama de Abreu M. Pressure support ventilation and biphasic positive airway pressure improve oxygenation by redistribution of pulmonary blood flow. Anesth Analg. 2009 Sep;109(3):856-65. doi: 10.1213/ane.0b013e3181aff245. PMID 19690258
- [Background] He H, Chi Y, Long Y, Yuan S, Zhang R, Yang Y, Frerichs I, Moller K, Fu F, Zhao Z. Three broad classifications of acute respiratory failure etiologies based on regional ventilation and perfusion by electrical impedance tomography: a hypothesis-generating study. Ann Intensive Care. 2021 Aug 28;11(1):134. doi: 10.1186/s13613-021-00921-6. PMID 34453622
- [Background] Spinelli E, Kircher M, Stender B, Ottaviani I, Basile MC, Marongiu I, Colussi G, Grasselli G, Pesenti A, Mauri T. Unmatched ventilation and perfusion measured by electrical impedance tomography predicts the outcome of ARDS. Crit Care. 2021 Jun 3;25(1):192. doi: 10.1186/s13054-021-03615-4. PMID 34082795
- [Background] Liu L, Xie J, Wang C, Zhao Z, Chong Y, Yuan X, Qiu H, Zhao M, Yang Y, Slutsky AS. Prone position improves lung ventilation-perfusion matching in non-intubated COVID-19 patients: a prospective physiologic study. Crit Care. 2022 Jun 29;26(1):193. doi: 10.1186/s13054-022-04069-y. No abstract available. PMID 35768877
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692